CLINICAL TRIAL: NCT07110935
Title: Efficacy of Treatment of Postpartum Anaemia With Intravenous Iron Versus Oral Iron
Brief Title: Efficacy of Treatment of Postpartum Anaemia With Intravenous Iron Versus Oral Iron in a Tertiary Hospital in South East, Nigeria.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Federal Teaching Hospital Abakaliki (Other Government)
Responsible Party: Principal Investigator, Assumpta Nnenna Nweke, Dr Assumpta Nnenna Nweke, Federal Teaching Hospital Abakaliki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMC/QEH/G.596/Vol.10/266
Record Dates: First submitted 2025-07-27; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Postpartum Anaemia
MeSH Terms: interventions — Iron

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One hundred and forty five women who picked "i" were assigned intravenous iron therapy group (Experimental)
  Interventions: Drug: intravenous iron
- One hundred and forty five women who picked "o" were assigned oral iron therapy group (Active Comparator)
  Interventions: Drug: oral iron

INTERVENTIONS:
Drug: intravenous iron — intravenous iron dextran
  Arms: One hundred and forty five women who picked "i" were assigned intravenous iron therapy group
Drug: oral iron — oral iron(ferrous Sulphate)
  Arms: One hundred and forty five women who picked "o" were assigned oral iron therapy group

SUMMARY:
Background:Anaemia is a condition of public health importance.Iron deficiency anaemia is the most common cause of anaemia in pregnancy.Postpartum anaemia poses a significant role for postpartum morbidity and mortality and should be treated.Postpartum iron deficiency anaemia warrants greater attention and higher quality of care.Oral iron treatment has been considered the standard of care.

However,parenteral iron treatment is expected to be advantageous in cases where oral iron therapy is not possible.As a result,there is increased interest in parenteral iron therapy.

Objectives:To determine the effect of treatment of postpartum anaemia with intravenous versus oral iron therapy at Federal Medical Centre,Umuahia.

Materials and Method:This study is a prospective randomized controlled study carried out in department of Obstetric and Gynaecology, Federal Medical Centre,Umuahia,the capital of Abia State,South-east, Nigeria. The study population comprised of postpartum women with mild to moderate anaemia within 48 hours of delivery who were randomized into two groups.One group will be given oral iron therapy and the other intravenous iron dextran.Response and comparative effects of treatment using either route of administration were assessed at 6 weeks postpartum.The biodata,obstetric characteristics and haemoglobin estimation of the respondents were recorded on a structured study proforma.The data obtained from the study was analyzed with the statistical package for the social sciences(SPSS) software.Continuous variables obtained from this study were expressed as mean and standard deviation while categorical variables were summarized using frequency and percentages.Association between categorical variables were done using chi square.P-value less than 0.05 was taken as significant.

ELIGIBILITY:
Inclusion Criteria:

* Women who have vaginal delivery of singleton baby and are seen within 48hours of childbirth
* Women with mild and moderate anaemia
* Women who gave their consent to participate in the study.

Exclusion Criteria:

* Women with severe anaemia
* Women with multiple pregnancy
* Women with genotype HbSS
* Women with HIV infection
* Women who delivered by caesarean section
* Women with co-morbidity like hypertensive disorders, renal pathology
* Women who decline consent after adequate counseling.
* Previous and current history of adverse reaction to iron dextran

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 290 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
Mean postpartum haematocrit | Six weeks
Mean hematocrit following treatment with iron dextran | Six weeks

SECONDARY OUTCOMES:
Incidence and patterns of postpartum anaemia | Six weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Federal Medical Centre , Umuahia, Umuahia, Abia State, Nigeria

IPD SHARING:
Plan to Share IPD: No